CLINICAL TRIAL: NCT01371799
Title: A Double Blind, Randomized, Placebo Controlled, Cross-over Study to Examine the Pharmacodynamic Effects of GSK1034702 on Neurophysiological Biomarkers of Cognition in Nicotine Abstained Otherwise Healthy Smokers
Brief Title: A Study to Examine the Pharmacodynamic Effects of GSK1034702 on Neurophysiological Biomarkers of Cognition in Nicotine Abstained Otherwise Healthy Smokers
Acronym: MAA113746
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 113746
Record Dates: First submitted 2011-04-14; First posted 2011-06-13 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Mental Disorders
Keywords: Schizophrenia
MeSH Terms: conditions — Mental Disorders; Schizophrenia | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study drug at 4mg (Experimental): GSK1034702 at 4mg
  Interventions: Drug: Drug
- Study drug at 8mg (Experimental): GSK1034702 at 8mg
  Interventions: Drug: Drug
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Drug

INTERVENTIONS:
Drug: Drug — Placebo
  Arms: Study drug at 4mg; Study drug at 8mg
Drug: Drug — 4mg and 8mg Study drug
  Arms: Placebo

SUMMARY:
This will be a double blind, randomised, placebo controlled, cross over study in which up to 20 otherwise healthy male nicotine abstinent smokers will be tested following 3 acute treatment conditions (placebo, 4 and 8mg of GSK1034702). Each subject will undergo screening assessments within 30 days prior to administration of the first dose of study medication. There will be 3 treatment sessions and dosing will be separated by a minimum 1 week washout period. There will be two testing days (day 1 and day 2) per treatment session. On each treatment session subjects will be admitted on day 1. On day 1, subjects will be administered placebo and approximately 3 hours later, there will be a Baseline EEG/ERP recording, neuropsychological (Cogstate battery) testing and mood/craving/dependence questionnaire assessments . Subjects will be allowed to smoke until approximately midnight on day 1. On day 2, subjects will undergo a pre-drug neuropsychological (Cogstate battery) testing and questionnaire assessments of mood/craving. This will be conducted approximately 1 hour prior to dosing. Subjects will be randomized to one of six treatment sequences. Post dose EEG/ERP recording, neuropsychological (Cogstate battery) testing and mood/craving measurements will be conducted between 3 and 6 hours post treatment to coincide with peak pharmacokinetic effects. This testing will be performed approximately at 12pm following at least 12hrs of nicotine abstinence. Blood samples will be collected at baseline (pre-drug) and following drug administration to quantify exposure levels.

ELIGIBILITY:
Inclusion Criteria A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Otherwise healthy smokers as determined by a responsible physician, based on a medical evaluation including own and familial medical history, physical examination, psychiatric history, psychiatric evaluation, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subjects must have QTc values within the normal range, i.e. QTcB or QTcF < 450 msec. The following normal ranges for blood pressure and heart rate are given as a guide: Systolic blood pressure ≥90 and ≤140 mmHg Diastolic blood pressure ≥60 and ≤90 mmHg Heart rate ≥50 and ≤90 bpm - Male subjects between 18 and 55 years of age.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1.1. This criterion must be followed from the time of the first dose of study medication until 3 months post-last dose.
* Subject is a smoker, i.e. on average smokes 10 or more cigarettes per day for at least 1 year prior to the screening visit. Urinary cotinine levels indicative of smoking at screening.
* Body weight > 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive).
* Subjects must have AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). Tests may be repeated once but must be within the above limits by the day one visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Current or past diagnosis of psychiatric disorder, as assessed by the MINI.
* Subjects, who in the investigator's judgement, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 6 months.
* Current or past diagnosis of cardiovascular disease including but not limited to hypertension, cardiac arrhythmias, personal or family history of long QT syndrome, cardiac conduction disorder and/or risk factors for coronary artery disease (i.e. family history in more than 2 first degree relatives) or other clinically significant cardiac disease
* Current or past diagnosis of cerebrovascular disease (e.g., stroke, transient ischemic attacks, aneurysms).
* Current or past diagnosis of autonomic dysfunction (e.g. prone to fainting, orthostatic hypotension). Current or past diagnosis of acute or chronic respiratory disease (excluding childhood asthma and allergic rhinitis) and/or abnormal spirometry for age, sex and height at screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a history of gastrointestinal bleeding and/or a history of peptic ulcer disease and/or presence of active gastrointestinal disease.
* Subjects with an unstable medical disorder or a disorder (including surgical interventions) that would likely interfere with the action, absorption, distribution, metabolism or excretion of GSK1034702, may pose a safety concern, or interfere with accurate assessment of safety.
* History of regular alcohol consumption within 6 months of the study defined as: For males: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to a half-pint (220 mL) of beer or 1 (125 mL) measure of spirits or 1 glass (125 mL) of wine.
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort and Gingko biloba) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice (and exotic citrus fruits, grapefruit hybrids or fruit juices) from 7 days prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-12-17 (Actual); Primary Completion 2010-06-18 (Actual); Study Completion 2010-06-18 (Actual)

PRIMARY OUTCOMES:
Measures will include changes in cognition measures of specific biomarkers | 12 months
  To investigate the effects of GSK1034702 on the mismatch negativity neurophysiologic marker of cognition.

SECONDARY OUTCOMES:
Measures will include changes in the neurophysiologic markers of cognition | 12 Months
  To investigate the effects of GSK1034702 on other neurophysiologic markers of cognition including, P50 suppression, P300, PPI and synchronized oscillations.
Measures of changes in cognition biomarkers vs. the stduy drug | 12 months
  To investigate the relationship between changes in the above neurophysiologic markers of cognitive function and drug exposure
Measures of cogstate tests of attention in tests mentioned To investigate the effects of GSK1034702 on Cogstate neuropsychologic tests of attention, working memory, learning and executive function | 12 months
  To investigate the effects of GSK1034702 on Cogstate neuropsychologic tests of attention, working memory, learning and executive function
Measures of difference between the tests in cogstate and the drug levels at different concentrations To investigate the relationship between changes in Cogstate behavioural task performance and drug exposure | 12 months
  To investigate the relationship between changes in Cogstate behavioural task performance and drug exposure
Safety measures and PK parameters and PK parameters will be measures, Vital signs, BP. To obtain further safety and PK information following oral administration of GSK1034702 to healthy subjects | 12 months
  To obtain further safety and PK information following oral administration of GSK1034702 to healthy subjects
Measures in modd/craving To investigate changes in mood/craving in the nicotine "on" state (baseline), following nicotine abstinence and following treatment | 12 months
  To investigate changes in mood/craving in the nicotine "on" state (baseline), following nicotine abstinence and following treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nathan PJ, Watson J, Lund J, Davies CH, Peters G, Dodds CM, Swirski B, Lawrence P, Bentley GD, O'Neill BV, Robertson J, Watson S, Jones GA, Maruff P, Croft RJ, Laruelle M, Bullmore ET. The potent M1 receptor allosteric agonist GSK1034702 improves episodic memory in humans in the nicotine abstinence model of cognitive dysfunction. Int J Neuropsychopharmacol. 2013 May;16(4):721-31. doi: 10.1017/S1461145712000752. Epub 2012 Aug 29. PMID 22932339
- [Background] te Beek ET, Hay JL, Bullman JN, Burgess C, Nahon KJ, Klaassen ES, Gray FA, van Gerven JM. Pharmacokinetics and central nervous system effects of the novel dual NK1 /NK3 receptor antagonist GSK1144814 in alcohol-intoxicated volunteers. Br J Clin Pharmacol. 2013 May;75(5):1328-39. doi: 10.1111/bcp.12004. PMID 23067311
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113746 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113746?search=study&study_ids=113746#rs
- Available data/document: Individual Participant Data Set: 113746 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113746 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113746 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113746 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113746 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113746 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register